CLINICAL TRIAL: NCT03060447
Title: A Phase 1b, Randomized, Double-Blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of GS-9620 in Antiretroviral Treated HIV-1 Infected Controllers
Brief Title: Study to Evaluate the Safety and Efficacy of Vesatolimod in Antiretroviral Treated Human Immunodeficiency Virus (HIV-1) Infected Controllers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-382-3961
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Results first posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-03

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — vesatolimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vesatolimod (Experimental): Participants in Period 1 will receive 10 doses of vesatolimod (4 mg to 8 mg) once every 14 days over a 20-week period along with their prescribed ART. Participants in Period 2 (ATI) will discontinue ART and vesatolimod and will be monitored for rebound in HIV-1 plasma viremia for 24 weeks. Participants who restart ART during Period 2 due to virologic rebound will complete the ART Re-Initiation Visits, and then Post-ART Re-suppression Visits monthly for 6 additional months. Participants who complete 24 Weeks of ATI without restarting ART will move onto Period 3 and have 2 options. They can remain off ART for up to an additional 24 weeks. Those who restart ART at the start of Period 3 will complete ART Re-initiation Visits and then Post-ART Re-suppression Visits monthly for 6 additional months.
  Interventions: Drug: Vesatolimod; Drug: ART
- Placebo (Experimental): Participants in Period 1 will receive 10 doses of placebo matched to vesatolimod once every 14 days over a 20-week period along with their prescribed ART. Participants in Period 2 (ATI) will discontinue ART and placebo and will be monitored for rebound in HIV-1 plasma viremia for 24 weeks. Participants who restart ART during Period 2 due to virologic rebound will complete the ART Re-Initiation Visits, and then Post-ART Re-suppression Visits monthly for 6 additional months. Participants who complete 24 Weeks of ATI without restarting ART will move onto Period 3 and have 2 options. They can remain off ART for up to an additional 24 weeks. Those who restart ART at the start of Period 3 will complete ART Re-initiation Visits and then Post-ART Re-suppression Visits monthly for 6 additional months.
  Interventions: Drug: Placebo; Drug: ART

INTERVENTIONS:
Drug: Vesatolimod — Tablets Administered orally
  Other Names: GS-9620
  Arms: Vesatolimod
Drug: Placebo — Tablets Administered orally
  Arms: Placebo
Drug: ART — ART regimens administered in accordance with their prescribing information. The following agents are allowed as part of the ART regimen: nucleoside reverse transcriptase inhibitors, raltegravir, dolutegravir (DTG), rilpivirine, and maraviroc.

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of a 10-dose regimen of vesatolimod in HIV-1 infected controllers on antiretroviral treatment (ART) and during analytical treatment interruption (ATI) following vesatolimod dosing.

ELIGIBILITY:
Key Inclusion Criteria:

* Plasma HIV-1 ribonucleic acid (RNA) levels < 50 copies/mL at screening
* Chronic HIV-1 infection (for ≥ 6 months) prior to ART initiation
* Pre-ART Plasma HIV-1 RNA set point between 50 and ≤ 5,000 copies/mL measured within two years prior to ART initiation
* On ART for ≥ 6 consecutive months prior to screening
* Documented plasma HIV-1 RNA < 50 copies/mL for ≥ 6 months preceding the screening visit (or undetectable HIV-1 RNA level according to the local assay being used if the limit of detection is ≥ 50 copies/mL). Unconfirmed virologic elevations of ≥ 50 copies/mL (transient detectable viremia, or "blip") prior to screening are acceptable.
* No documented history of resistance to any components of the current ART regimen
* Availability of a fully active alternative ART regimen, in the opinion of the Investigator, in the event of discontinuation of the current ART regimen with development of resistance.
* Hemoglobin ≥ 11.5 g/dL (males) or ≥ 11 g/dL (females)
* White Blood Cells ≥ 2,500 cells/μL
* Platelets ≥ 125,000/mL
* Absolute Neutrophil Counts ≥ 1000 cells/μL
* Cluster of Differentiation 4 (CD4)+ count ≥ 500 cells/μL
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST) or bilirubin ≤ 2 × upper limit of normal (ULN)
* Estimated glomerular filtration rate ≥ 60 mL/min
* No autoimmune disease requiring on-going immunosuppression
* No evidence of current hepatitis B virus (HBV) infection
* No evidence of current hepatitis C virus (HCV) infection (positive anti-HCV antibody and negative HCV polymerase chain reaction (PCR) results are acceptable)
* No documented history of pre-ART CD4 nadir < 200 cells/μL (unknown pre-ART CD4 nadir is acceptable)
* No history of opportunistic illness indicative of stage 3 HIV
* No acute febrile illness within 35 days prior to Pre-Baseline/ Day -13

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (6):
- United States (6):
  - Mills Clinical Research, Los Angeles, California
  - Zuckerberg San Francisco General, San Francisco, California
  - Midway Immunology & Research Center, Ft. Pierce, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Central Texas Clinical Research, Austin, Texas
  - Peter Shalit, MD, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] SenGupta D, Ramgopal M, Brinson C, DeJesus E, Mills A, Shalit P, et al. Safety and Analytic Treatment Interruption Outcomes of Vesatolimod in HIV Controllers. Oral Presentation at CROI 2020, Boston, USA. Abstract 3982.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 09 May 2017. The last study visit occurred on 13 February 2020.
Pre-assignment Details: 31 participants were screened.
Groups:
- Vesatolimod: Participants in Period 1 received 10 doses of vesatolimod (4 mg to 8 mg) tablets once every 14 days over a 20-week period along with their prescribed antiretroviral treatment (ART). Participants in Period 2 (ATI) discontinued ART and vesatolimod and were monitored for rebound in HIV-1 plasma viremia for 24 weeks. Participants who restarted ART during Period 2 due to virologic rebound completed the ART Re-Initiation Visits, and then Post-ART Re-suppression Visits monthly for 6 additional months. Participants who completed 24 Weeks of ATI without restarting ART moved onto Period 3 and had 2 options. They remained off ART for up to an additional 24 weeks. Those who restarted ART at the start of Period 3 completed ART Re-initiation Visits and then Post-ART Re-suppression Visits monthly for 6 additional months.
- Placebo: Participants in Period 1 received 10 doses of placebo matched to vesatolimod tablets once every 14 days over a 20-week period along with their prescribed ART. Participants in Period 2 (ATI) discontinued ART and placebo and were monitored for rebound in HIV-1 plasma viremia for 24 weeks. Participants who restarted ART during Period 2 due to virologic rebound completed the ART Re-Initiation Visits, and then Post-ART Re-suppression Visits monthly for 6 additional months. Participants who completed 24 Weeks of ATI without restarting ART moved onto Period 3 and had 2 options. They remained off ART for up to an additional 24 weeks. Those who restarted ART at the start of Period 3 completed ART Re-initiation Visits and then Post-ART Re-suppression Visits monthly for 6 additional months.
Period: Overall Study
Arm/Group | Vesatolimod | Placebo
Started | 17 | 8
Completed | 15 | 8
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who were randomized and received at least 1 dose of study drug.
Groups:
- Vesatolimod: Participants in Period 1 received 10 doses of vesatolimod (4 mg to 8 mg) tablets once every 14 days over a 20-week period along with their prescribed ART. Participants in Period 2 (ATI) discontinued ART and vesatolimod and were monitored for rebound in HIV-1 plasma viremia for 24 weeks. Participants who restarted ART during Period 2 due to virologic rebound completed the ART Re-Initiation Visits, and then Post-ART Re-suppression Visits monthly for 6 additional months. Participants who completed 24 Weeks of ATI without restarting ART moved onto Period 3 and had 2 options. They remained off ART for up to an additional 24 weeks. Those who restarted ART at the start of Period 3 completed ART Re-initiation Visits and then Post-ART Re-suppression Visits monthly for 6 additional months.
- Total: Total of all reporting groups
Arm/Group | Vesatolimod | Placebo | Total
Number analyzed (Participants) | 17 | 8 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (11.4) | 42 (9.4) | 46 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 13 | 8 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 17 | 7 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 11 | 6 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 1.30 (0.108) | 1.28 (0.000) | 1.30 (0.089)
HIV-1 RNA Category [Count of Participants; unit: Participants]
  < 50 copies/mL | 16 | 8 | 24
  ≥ 50 copies/mL | 1 | 0 | 1
Pre-ART Plasma Viral Set-point [Mean (Standard Deviation); unit: log10 copies/mL] | 3.15 (0.275) | 3.08 (0.469) | 3.13 (0.340)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Treatment Emergent Serious Adverse Events (TESAEs) and Treatment Emergent Adverse Events (TEAEs)
Description: AE was any untoward medical occurrence in a clinical study participant administered a medicinal product (MP), which did not necessarily had a causal relationship with treatment. AE was therefore any unfavorable and/or unintended sign, symptom, or disease temporally associated with use of MP, whether or not considered related to MP. TEAEs: AE with an onset date on or after the study drug start date and no later than 30 days after study drug stop date; or any AE leading to study drug discontinuation. TESAEs: event that resulted in following: death; life-threatening situation; in-patient hospitalization or prolongation of existing hospitalization; persistent or significant disability or incapacity; congenital anomaly or birth defect; medically important event or reaction: such events might not have been immediately life-threatening or resulted in death or hospitalization but may jeopardize participant or may require intervention to prevent one of the other outcomes constituting SAEs.
Time Frame: From first dose up to 30 days after permanent discontinuation of study drug (assessed maximum up to 33 months and 5 days)
Population: The Safety Analysis Set included all participants who were randomized and received at least 1 dose of study drug. Per planned analysis, this outcome measure was analyzed by vesatolimod dose level and placebo.
Measure: Number; unit: percentage of participants
Groups:
- Vesatolimod 4 mg: Participants in Period 1 received 10 doses of vesatolimod 4 mg tablets once every 14 days over a 20-week period along with their prescribed ART. Participants in Period 2 (ATI) discontinued ART and vesatolimod and were monitored for rebound in HIV-1 plasma viremia for 24 weeks. Participants who restarted ART during Period 2 due to virologic rebound completed the ART Re-Initiation Visits, and then Post-ART Re-suppression Visits monthly for 6 additional months. Participants who completed 24 Weeks of ATI without restarting ART moved onto Period 3 and had 2 options. They remained off ART for up to an additional 24 weeks. Those who restarted ART at the start of Period 3 completed ART Re-initiation Visits and then Post-ART Re-suppression Visits monthly for 6 additional months.
- Vesatolimod 4/6 mg: Participants in Period 1 received 10 doses of vesatolimod 4 mg or 6 mg tablets once every 14 days over a 20-week period along with their prescribed ART. Participants in Period 2 (ATI) discontinued ART and vesatolimod and were monitored for rebound in HIV-1 plasma viremia for 24 weeks. Participants who restarted ART during Period 2 due to virologic rebound completed the ART Re-Initiation Visits, and then Post-ART Re-suppression Visits monthly for 6 additional months. Participants who completed 24 Weeks of ATI without restarting ART moved onto Period 3 and had 2 options. They remained off ART for up to an additional 24 weeks. Those who restarted ART at the start of Period 3 completed ART Re-initiation Visits and then Post-ART Re-suppression Visits monthly for 6 additional months.
- Vesatolimod 6 mg: Participants in Period 1 received 10 doses of vesatolimod 6 mg tablets once every 14 days over a 20-week period along with their prescribed ART. Participants in Period 2 (ATI) discontinued ART and vesatolimod and were monitored for rebound in HIV-1 plasma viremia for 24 weeks. Participants who restarted ART during Period 2 due to virologic rebound completed the ART Re-Initiation Visits, and then Post-ART Re-suppression Visits monthly for 6 additional months. Participants who completed 24 Weeks of ATI without restarting ART moved onto Period 3 and had 2 options. They remained off ART for up to an additional 24 weeks. Those who restarted ART at the start of Period 3 completed ART Re-initiation Visits and then Post-ART Re-suppression Visits monthly for 6 additional months.
- Vesatolimod 6/8 mg: Participants in Period 1 received 10 doses of vesatolimod 6 mg or 8 mg tablets once every 14 days over a 20-week period along with their prescribed ART. Participants in Period 2 (ATI) discontinued ART and vesatolimod and were monitored for rebound in HIV-1 plasma viremia for 24 weeks. Participants who restarted ART during Period 2 due to virologic rebound completed the ART Re-Initiation Visits, and then Post-ART Re-suppression Visits monthly for 6 additional months. Participants who completed 24 Weeks of ATI without restarting ART moved onto Period 3 and had 2 options. They remained off ART for up to an additional 24 weeks. Those who restarted ART at the start of Period 3 completed ART Re-initiation Visits and then Post-ART Re-suppression Visits monthly for 6 additional months.
- Vesatolimod 8 mg: Participants in Period 1 received 10 doses of vesatolimod 8 mg tablets once every 14 days over a 20-week period along with their prescribed ART. Participants in Period 2 (ATI) discontinued ART and vesatolimod and were monitored for rebound in HIV-1 plasma viremia for 24 weeks. Participants who restarted ART during Period 2 due to virologic rebound completed the ART Re-Initiation Visits, and then Post-ART Re-suppression Visits monthly for 6 additional months. Participants who completed 24 Weeks of ATI without restarting ART moved onto Period 3 and had 2 options. They remained off ART for up to an additional 24 weeks. Those who restarted ART at the start of Period 3 completed ART Re-initiation Visits and then Post-ART Re-suppression Visits monthly for 6 additional months.
Arm/Group | Vesatolimod 4 mg | Vesatolimod 4/6 mg | Vesatolimod 6 mg | Vesatolimod 6/8 mg | Vesatolimod 8 mg | Placebo
Number analyzed (Participants) | 2 | 4 | 5 | 3 | 3 | 8
percentage of participants
  TESAEs | 0 | 0 | 0 | 33.3 | 0 | 0
  TEAEs | 100.00 | 75.00 | 100.00 | 100.00 | 100.00 | 75.00

2. Secondary Outcome: Change From Baseline in Plasma Log 10 HIV-1 RNA by Taqman 2.0
Description: Plasma log 10 HIV-1 RNA was measured using Taqman version 2.0 assay with limit of quantification of 20 copies/mL.
Time Frame: Baseline and Dose 1: Days 2,8; Dose 2: Days 1,8; Dose 3: Days 1,8; Dose 4: Days 1,2,4,8; Dose 5: Day 1,8; Dose 6: Days 1,4,8; Dose 7: Days 1,8; Dose 8: Days 1,8; Dose 9: Days 1,8; Dose 10: Days 1,2,4,8,14
Population: Participants in the Full Analysis Set (included all participants who were randomized into the study and received at least one dose of study drug) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Vesatolimod | Placebo
Number analyzed (Participants) | 17 | 8
Log10 copies/mL
  Change at Dose 1: Day 2 | -0.01 (0.027) | 0.00 (0.000)
  Change at Dose 1: Day 8: number analyzed (Participants) | 16 | 8
  Change at Dose 1: Day 8 | 0.05 (0.212) | 0.00 (0.000)
  Change at Dose 2: Day 1: number analyzed (Participants) | 16 | 8
  Change at Dose 2: Day 1 | 0.09 (0.372) | 0.00 (0.000)
  Change at Dose 2: Day 8: number analyzed (Participants) | 16 | 8
  Change at Dose 2: Day 8 | -0.03 (0.111) | 0.00 (0.000)
  Change at Dose 3: Day 1: number analyzed (Participants) | 16 | 8
  Change at Dose 3: Day 1 | -0.03 (0.111) | 0.00 (0.000)
  Change at Dose 3: Day 8: number analyzed (Participants) | 16 | 7
  Change at Dose 3: Day 8 | -0.03 (0.111) | 0.00 (0.000)
  Change at Dose 4: Day 1: number analyzed (Participants) | 16 | 8
  Change at Dose 4: Day 1 | -0.03 (0.111) | 0.00 (0.000)
  Change at Dose 4: Day 2: number analyzed (Participants) | 15 | 8
  Change at Dose 4: Day 2 | -0.03 (0.115) | 0.00 (0.000)
  Change at Dose 4: Day 4: number analyzed (Participants) | 15 | 8
  Change at Dose 4: Day 4 | -0.03 (0.115) | 0.00 (0.000)
  Change at Dose 4: Day 8: number analyzed (Participants) | 16 | 6
  Change at Dose 4: Day 8 | -0.03 (0.111) | 0.00 (0.000)
  Change at Dose 5: Day 1: number analyzed (Participants) | 16 | 8
  Change at Dose 5: Day 1 | -0.03 (0.111) | 0.00 (0.000)
  Change at Dose 5: Day 8: number analyzed (Participants) | 15 | 8
  Change at Dose 5: Day 8 | -0.03 (0.115) | 0.00 (0.000)
  Change at Dose 6: Day 1: number analyzed (Participants) | 15 | 8
  Change at Dose 6: Day 1 | -0.03 (0.115) | 0.00 (0.000)
  Change at Dose 6: Day 4: number analyzed (Participants) | 15 | 8
  Change at Dose 6: Day 4 | -0.03 (0.115) | 0.00 (0.000)
  Change at Dose 6: Day 8: number analyzed (Participants) | 15 | 8
  Change at Dose 6: Day 8 | -0.03 (0.115) | 0.00 (0.000)
  Change at Dose 7: Day 1: number analyzed (Participants) | 15 | 8
  Change at Dose 7: Day 1 | -0.03 (0.115) | 0.00 (0.000)
  Change at Dose 7: Day 8: number analyzed (Participants) | 15 | 8
  Change at Dose 7: Day 8 | -0.03 (0.115) | 0.00 (0.000)
  Change at Dose 8: Day 1: number analyzed (Participants) | 15 | 8
  Change at Dose 8: Day 1 | -0.03 (0.115) | 0.00 (0.000)
  Change at Dose 8: Day 8: number analyzed (Participants) | 15 | 8
  Change at Dose 8: Day 8 | -0.03 (0.115) | 0.00 (0.000)
  Change at Dose 9: Day 1: number analyzed (Participants) | 15 | 8
  Change at Dose 9: Day 1 | -0.03 (0.115) | 0.00 (0.000)
  Change at Dose 9: Day 8: number analyzed (Participants) | 14 | 8
  Change at Dose 9: Day 8 | 0.00 (0.000) | 0.00 (0.000)
  Change at Dose 10: Day 1: number analyzed (Participants) | 15 | 8
  Change at Dose 10: Day 1 | -0.03 (0.115) | 0.00 (0.000)
  Change at Dose 10: Day 2: number analyzed (Participants) | 15 | 8
  Change at Dose 10: Day 2 | -0.03 (0.115) | 0.00 (0.000)
  Change at Dose 10: Day 4: number analyzed (Participants) | 15 | 8
  Change at Dose 10: Day 4 | -0.03 (0.115) | 0.00 (0.000)
  Change at Dose 10: Day 8: number analyzed (Participants) | 15 | 8
  Change at Dose 10: Day 8 | -0.03 (0.115) | 0.00 (0.000)
  Change at Dose 10: Day 14: number analyzed (Participants) | 15 | 8
  Change at Dose 10: Day 14 | -0.03 (0.115) | 0.00 (0.000)
Statistical Analysis 1: Comparison: Vesatolimod vs Placebo; Dose 1: Day 2; Test type: Superiority; p = 0.55, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 2: Comparison: Vesatolimod vs Placebo; Dose 1: Day 8; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 3: Comparison: Vesatolimod vs Placebo; Dose 2: Day 1; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 4: Comparison: Vesatolimod vs Placebo; Dose 2: Day 8; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 5: Comparison: Vesatolimod vs Placebo; Dose 3: Day 1; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 6: Comparison: Vesatolimod vs Placebo; Dose 3: Day 8; Test type: Superiority; p = 0.57, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 7: Comparison: Vesatolimod vs Placebo; Dose 4: Day 1; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 8: Comparison: Vesatolimod vs Placebo; Dose 4: Day 2; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 9: Comparison: Vesatolimod vs Placebo; Dose 4: Day 4; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 10: Comparison: Vesatolimod vs Placebo; Dose 4: Day 8; Test type: Superiority; p = 0.61, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 11: Comparison: Vesatolimod vs Placebo; Dose 5: Day 1; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 12: Comparison: Vesatolimod vs Placebo; Dose 5: Day 8; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 13: Comparison: Vesatolimod vs Placebo; Dose 6: Day 1; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 14: Comparison: Vesatolimod vs Placebo; Dose 6: Day 4; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 15: Comparison: Vesatolimod vs Placebo; Dose 6: Day 8; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 16: Comparison: Vesatolimod vs Placebo; Dose 7: Day 1; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 17: Comparison: Vesatolimod vs Placebo; Dose 7 - Day 8; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 18: Comparison: Vesatolimod vs Placebo; Dose 8: Day 1; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 19: Comparison: Vesatolimod vs Placebo; Dose 8: Day 8; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 20: Comparison: Vesatolimod vs Placebo; Dose 9: Day 1; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 21: Comparison: Vesatolimod vs Placebo; Dose 9: Day 8; Test type: Superiority; p = 1.00, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 22: Comparison: Vesatolimod vs Placebo; Dose 10: Day 1; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 23: Comparison: Vesatolimod vs Placebo; Dose 10: Day 2; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 24: Comparison: Vesatolimod vs Placebo; Dose 10: Day 4; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 25: Comparison: Vesatolimod vs Placebo; Dose 10: Day 8; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 26: Comparison: Vesatolimod vs Placebo; Dose 10: Day 14; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests

3. Secondary Outcome: Time to Virologic Rebound
Description: Time to virologic rebound was analyzed using the Kaplan-Meier method at two cut-off values; ≥ 50 copies/mL and ≥ 200 copies/mL. Virologic rebound at ≥ 50 copies/mL was defined as 2 consecutive HIV-1 RNA measurements ≥ 50 copies/mL. Virologic rebound at ≥ 200 copies/mL was defined as 2 consecutive HIV-1 RNA measurements ≥ 200 copies/mL. The date of rebound was the first time HIV-1 RNA measurement ≥ 50 copies/mL or ≥ 200 respectively.
Time Frame: From Day 1 (Period 1) up to 24 weeks of Period 2 plus 6 months following virologic re-suppression on ART, an average of 17 months
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Vesatolimod | Placebo
Number analyzed (Participants) | 15 | 8
weeks
  ≥ 50 Copies/mL | 4.3 [3.1 to 6.1] | 4.0 [3.0 to 4.2]
  ≥ 200 Copies/mL | 5.1 [4.1 to 6.3] | 4.1 [3.8 to 4.6]
Statistical Analysis 1: Comparison: Vesatolimod vs Placebo; ≥ 50 Copies/mL; Test type: Superiority; p = 0.035, Log Rank; P-value between treatment groups was based on log-rank test
Statistical Analysis 2: Comparison: Vesatolimod vs Placebo; ≥ 200 Copies/mL; Test type: Superiority; p = 0.024, Log Rank; P-value between treatment groups was based on log-rank test

4. Secondary Outcome: Peak HIV-1 Viral Load During Period 2
Description: For participants who did not restart ART, the maximum value of HIV-1 RNA measurements during ATI was used as the peak value and for participants who restarted ART, the maximum value of HIV-1 RNA measurements during ATI before the restart of ART was used as the peak value.
Time Frame: From Week 1 up to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: Log10 copies/mL
Arm/Group | Vesatolimod | Placebo
Number analyzed (Participants) | 15 | 8
Log10 copies/mL | 4.21 [3.39 to 4.88] | 3.97 [3.29 to 4.32]
Statistical Analysis 1: Comparison: Vesatolimod vs Placebo; Test type: Superiority; p = 0.67, Wilcoxon (Mann-Whitney); P-values between treatment groups were based on Wilcoxon rank sum test

5. Secondary Outcome: Change in Plasma Viral Load Set-Point Following ATI
Description: Plasma viral load set-point values were calculated at pre-ART stage and following ATI. Change in plasma viral load set-point following ATI = viral set-point following ATI minus pre-ART set point. The plasma viral set-point following ATI was calculated as the geometric mean of all the HIV-1 RNA measurements between a start date and an end date. The start date and end date was provided by clinical based on blinded individual participant's data review.
Time Frame: Pre-ART (Initial Screening Visit) and 24 weeks plus 6 months following virologic re-suppression on ART (maximum 33 months and 5 days)
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: Log10 copies/mL
Arm/Group | Vesatolimod | Placebo
Number analyzed (Participants) | 15 | 7
Log10 copies/mL | -0.37 [-0.59 to -0.05] | -0.28 [-0.56 to 0.17]
Statistical Analysis 1: Comparison: Vesatolimod vs Placebo; Test type: Superiority; p = 0.78, Wilcoxon (Mann-Whitney); P-values between treatment groups were based on Wilcoxon rank sum test

6. Secondary Outcome: Change From Baseline in Levels of Serum Cytokines
Description: Following Serum Cytokines Levels were evaluated: interferon-a (IFN-a), interleukin-1 receptor antagonist (IL-1RA), inducible protein-10 (IP-10) and inducible T cell alpha chemoattractant (ITAC).
Time Frame: Baseline and Dose 1: Day 2,8; Dose 4: Days 1,2,8; Dose 10: Days 1,2,8; ATI Remission Visit (12 weeks post ATI Visit: evaluated at maximum of 24 weeks); Early study drug discontinuation (7 days post- last ATI visit at Week 24)
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Vesatolimod | Placebo
Number analyzed (Participants) | 17 | 8
pg/mL
  IFN-a, Baseline | 0.02 (0.036) | 0.05 (0.075)
  IFN-a,Change at Dose 1: Day 2 | 0.41 (0.834) | -0.01 (0.073)
  IFN-a,Change at Dose 1: Day 8: number analyzed (Participants) | 16 | 8
  IFN-a,Change at Dose 1: Day 8 | 0.14 (0.447) | 0.04 (0.129)
  IFN-a,Change at Dose 4: Day 1: number analyzed (Participants) | 16 | 8
  IFN-a,Change at Dose 4: Day 1 | -0.01 (0.030) | 0.10 (0.358)
  IFN-a,Change at Dose 4: Day 2: number analyzed (Participants) | 16 | 8
  IFN-a,Change at Dose 4: Day 2 | 0.75 (2.361) | -0.01 (0.065)
  IFN-a,Change at Dose 4: Day 8: number analyzed (Participants) | 16 | 6
  IFN-a,Change at Dose 4: Day 8 | 0.01 (0.064) | -0.03 (0.077)
  IFN-a,Change at Dose 10: Day 1: number analyzed (Participants) | 15 | 8
  IFN-a,Change at Dose 10: Day 1 | -0.01 (0.031) | -0.03 (0.056)
  IFN-a,Change at Dose 10: Day 2: number analyzed (Participants) | 15 | 8
  IFN-a,Change at Dose 10: Day 2 | 0.51 (1.028) | -0.02 (0.055)
  IFN-a,Change at Dose 10: Day 8: number analyzed (Participants) | 15 | 8
  IFN-a,Change at Dose 10: Day 8 | 0.01 (0.072) | -0.04 (0.065)
  IFN-a,Change at ATI Remission Visit: number analyzed (Participants) | 4 | 3
  IFN-a,Change at ATI Remission Visit | -0.03 (0.059) | 0.17 (0.301)
  IFN-a,Change at Early study drug discontinuation: number analyzed (Participants) | 1 | 0
  IFN-a,Change at Early study drug discontinuation | 0.00 |
  IL-1RA, Baseline: number analyzed (Participants) | 15 | 8
  IL-1RA, Baseline | 2346.1 (3743.44) | 882.9 (306.75)
  IL-1RA,Change at Dose 1: Day 2: number analyzed (Participants) | 14 | 8
  IL-1RA,Change at Dose 1: Day 2 | 2797.6 (2908.21) | 94.8 (190.53)
  IL-1RA,Change at Dose 1: Day 8: number analyzed (Participants) | 12 | 6
  IL-1RA,Change at Dose 1: Day 8 | -326.9 (914.43) | 1004.9 (2432.36)
  IL-1RA,Change at Dose 4: Day 1: number analyzed (Participants) | 13 | 7
  IL-1RA,Change at Dose 4: Day 1 | 390.4 (856.29) | 42.2 (227.90)
  IL-1RA,Change at Dose 4: Day 2: number analyzed (Participants) | 13 | 7
  IL-1RA,Change at Dose 4: Day 2 | 5140.4 (8692.35) | 186.4 (449.94)
  IL-1RA,Change at Dose 4: Day 8: number analyzed (Participants) | 14 | 5
  IL-1RA,Change at Dose 4: Day 8 | -63.9 (1749.75) | -143.5 (226.83)
  IL-1RA,Change at Dose 10: Day 1: number analyzed (Participants) | 12 | 7
  IL-1RA,Change at Dose 10: Day 1 | -160.9 (1229.91) | 563.9 (1201.78)
  IL-1RA,Change at Dose 10: Day 2: number analyzed (Participants) | 13 | 8
  IL-1RA,Change at Dose 10: Day 2 | 3790.2 (6401.27) | 14.1 (467.90)
  IL-1RA,Change at Dose 10: Day 8: number analyzed (Participants) | 12 | 7
  IL-1RA,Change at Dose 10: Day 8 | -77.6 (521.52) | -13.9 (308.80)
  IL-1RA,Change at ATI Remission Visit: number analyzed (Participants) | 3 | 2
  IL-1RA,Change at ATI Remission Visit | -161.7 (1030.42) | 491.1 (306.12)
  IL-1RA,Change at Early study drug discontinuation: number analyzed (Participants) | 1 | 0
  IL-1RA,Change at Early study drug discontinuation | 222.4 |
  IP-10, Baseline | 161.0 (82.04) | 178.5 (103.50)
  IP-10, Change at Dose 1: Day 2 | 554.1 (693.55) | -23.9 (52.24)
  IP-10,Change at Dose 1: Day 8: number analyzed (Participants) | 16 | 8
  IP-10,Change at Dose 1: Day 8 | 38.8 (126.82) | 34.5 (182.93)
  IP-10,Change at Dose 4: Day 1: number analyzed (Participants) | 16 | 8
  IP-10,Change at Dose 4: Day 1 | 27.8 (71.62) | -25.3 (46.15)
  IP-10,Change at Dose 4: Day 2: number analyzed (Participants) | 16 | 8
  IP-10,Change at Dose 4: Day 2 | 337.9 (487.83) | -13.8 (78.10)
  IP-10,Change at Dose 4: Day 8: number analyzed (Participants) | 16 | 6
  IP-10,Change at Dose 4: Day 8 | 23.4 (58.50) | -59.0 (58.04)
  IP-10,Change at Dose 10: Day 1: number analyzed (Participants) | 15 | 8
  IP-10,Change at Dose 10: Day 1 | 19.1 (44.13) | -22.8 (54.29)
  IP-10,Change at Dose 10: Day 2: number analyzed (Participants) | 15 | 8
  IP-10,Change at Dose 10: Day 2 | 554.6 (893.70) | -17.5 (50.94)
  IP-10, Change at Dose 10: Day 8: number analyzed (Participants) | 15 | 8
  IP-10, Change at Dose 10: Day 8 | 18.1 (82.14) | -51.1 (57.23)
  IP-10,Change at ATI Remission: number analyzed (Participants) | 4 | 3
  IP-10,Change at ATI Remission | 47.5 (48.42) | 26.2 (92.41)
  IP-10,Change at Early Study Drug Discontinuation: number analyzed (Participants) | 1 | 0
  IP-10,Change at Early Study Drug Discontinuation | 0.7 |
  ITAC, Baseline | 71.8 (108.10) | 206.3 (329.55)
  ITAC, Change at Dose 1: Day 2 | 50.4 (80.46) | -13.9 (42.68)
  ITAC,Change at Dose 1: Day 8: number analyzed (Participants) | 16 | 8
  ITAC,Change at Dose 1: Day 8 | 11.5 (34.78) | -10.4 (44.02)
  ITAC, Change at Dose 4: Day 1: number analyzed (Participants) | 16 | 8
  ITAC, Change at Dose 4: Day 1 | 8.0 (25.97) | -25.4 (65.76)
  ITAC,Change at Dose 4: Day 2: number analyzed (Participants) | 16 | 8
  ITAC,Change at Dose 4: Day 2 | 48.0 (78.14) | -8.9 (33.81)
  ITAC, Change at Dose 4: Day 8: number analyzed (Participants) | 16 | 6
  ITAC, Change at Dose 4: Day 8 | 2.0 (24.20) | 5.0 (27.98)
  ITAC,Change at Dose 10: Day 1: number analyzed (Participants) | 15 | 8
  ITAC,Change at Dose 10: Day 1 | -1.6 (19.11) | -8.4 (33.91)
  ITAC,Change at Dose 10: Day 2: number analyzed (Participants) | 15 | 8
  ITAC,Change at Dose 10: Day 2 | 69.1 (181.55) | -1.0 (27.68)
  ITAC,Change at Dose 10: Day 8: number analyzed (Participants) | 15 | 8
  ITAC,Change at Dose 10: Day 8 | 2.2 (12.19) | -7.4 (22.50)
  ITAC,Change at ATI Remission: number analyzed (Participants) | 4 | 3
  ITAC,Change at ATI Remission | 19.1 (20.44) | 39.6 (88.54)
  ITAC,Change at Early Study Drug Discontinuation: number analyzed (Participants) | 1 | 0
  ITAC,Change at Early Study Drug Discontinuation | 31.2 |
Statistical Analysis 1: Comparison: Vesatolimod vs Placebo; IFN-a, Baseline; Test type: Superiority; p = 0.34, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 2: Comparison: Vesatolimod vs Placebo; IFN-a, Dose 1: Day 2; Test type: Superiority; p = 0.11, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 3: Comparison: Vesatolimod vs Placebo; IFN-a, Dose 1: Day 8; Test type: Superiority; p = 0.81, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 4: Comparison: Vesatolimod vs Placebo; IFN-a, Dose 4: Day 1; Test type: Superiority; p = 0.83, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 5: Comparison: Vesatolimod vs Placebo; IFN-a, Dose 4: Day 2; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 6: Comparison: Vesatolimod vs Placebo; IFN-a, Dose 4: Day 8; Test type: Superiority; p = 0.45, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 7: Comparison: Vesatolimod vs Placebo; IFN-a, Dose 10: Day 1; Test type: Superiority; p = 0.25, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 8: Comparison: Vesatolimod vs Placebo; IFN-a, Dose 10: Day 2; Test type: Superiority; p = 0.053, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 9: Comparison: Vesatolimod vs Placebo; IFN-a, Dose 10: Day 8; Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 10: Comparison: Vesatolimod vs Placebo; IFN-a, ATI Remission Visit; Test type: Superiority; p = 0.27, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 11: Comparison: Vesatolimod vs Placebo; IL-1RA, Baseline; Test type: Superiority; p = 0.35, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 12: Comparison: Vesatolimod vs Placebo; IL-1RA, Dose 1: Day 2; Test type: Superiority; p = 0.013, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 13: Comparison: Vesatolimod vs Placebo; IL-1RA, Dose 1: Day 8; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 14: Comparison: Vesatolimod vs Placebo; IL-1RA, Dose 4: Day 1; Test type: Superiority; p = 0.30, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 15: Comparison: Vesatolimod; IL-1RA, Dose 4: Day 2; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 16: Comparison: Vesatolimod vs Placebo; IL-1RA, Dose 4: Day 8; Test type: Superiority; p = 0.49, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 17: Comparison: Vesatolimod vs Placebo; IL-1RA, Dose 10: Day 1; Test type: Superiority; p = 0.25, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 18: Comparison: Vesatolimod vs Placebo; IL-1RA, Dose 10: Day 2; Test type: Superiority; p = 0.055, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 19: Comparison: Vesatolimod vs Placebo; IL-1RA, Dose 10: Day 8; Test type: Superiority; p = 0.90, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 20: Comparison: Vesatolimod vs Placebo; IL-1RA, ATI Remission Visit; Test type: Superiority; p = 0.39, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 21: Comparison: Vesatolimod vs Placebo; IP-10, Baseline; Test type: Superiority; p = 0.75, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 22: Comparison: Vesatolimod vs Placebo; IP-10, Dose 1: Day 2; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 23: Comparison: Vesatolimod vs Placebo; IP-10, Dose 1: Day 8; Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 24: Comparison: Vesatolimod vs Placebo; IP-10, Dose 4: Day 1; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 25: Comparison: Vesatolimod vs Placebo; IP-10, Dose 4: Day 2; Test type: Superiority; p = 0.018, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 26: Comparison: Vesatolimod vs Placebo; IP-10, Dose 4: Day 8; Test type: Superiority; p = 0.030, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 27: Comparison: Vesatolimod vs Placebo; IP-10, Dose 10: Day 1; Test type: Superiority; p = 0.087, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 28: Comparison: Vesatolimod vs Placebo; IP-10, Dose 10: Day 2; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 29: Comparison: Vesatolimod vs Placebo; IP-10, Dose 10: Day 8; Test type: Superiority; p = 0.066, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 30: Comparison: Vesatolimod vs Placebo; IP-10, ATI Remission; Test type: Superiority; p = 0.86, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 31: Comparison: Vesatolimod vs Placebo; ITAC, Baseline; Test type: Superiority; p = 0.19, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 32: Comparison: Vesatolimod vs Placebo; ITAC, Dose 1: Day 2; Test type: Superiority; p = 0.021, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 33: Comparison: Vesatolimod vs Placebo; ITAC, Dose 1: Day 8; Test type: Superiority; p = 0.31, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 34: Comparison: Vesatolimod vs Placebo; ITAC, Dose 4: Day 1; Test type: Superiority; p = 0.10, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 35: Comparison: Vesatolimod vs Placebo; ITAC, Dose 4: Day 2; Test type: Superiority; p = 0.018, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 36: Comparison: Vesatolimod vs Placebo; ITAC, Dose 4: Day 8; Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 37: Comparison: Vesatolimod vs Placebo; ITAC, Dose 10: Day 1; Test type: Superiority; p = 0.46, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 38: Comparison: Vesatolimod vs Placebo; ITAC, Dose 10: Day 2; Test type: Superiority; p = 0.21, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 39: Comparison: Vesatolimod vs Placebo; ITAC, Dose 10: Day 8; Test type: Superiority; p = 0.67, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 40: Comparison: Vesatolimod vs Placebo; ITAC, ATI Remission; Test type: Superiority; p = 0.60, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests

7. Secondary Outcome: Fold Change in Messenger Ribonucleic Acid (mRNA) of Interferon-Stimulated Genes (ISGs) in Whole Blood
Description: Following ISGs Levels were evaluated: Interferon-stimulated Gene 15 (ISG15), Oligoadenylate synthase-1 (OAS-1), and interferon-induced guanosine triphosphate-binding protein MX1. Fold change was calculated as postbaseline value divided by baseline value.
Time Frame: Baseline and Dose 1: Day 2; Dose 4: Days 1,2; Dose 10: Day 1,2; Early Study Drug Discontinuation (7 days post- last ATI visit at Week 24)
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Vesatolimod | Placebo
Number analyzed (Participants) | 17 | 8
fold change
  ISG15, Dose 1: Day 2 | 19.53 (15.548) | 1.06 (0.320)
  ISG15, Dose 4: Day 1: number analyzed (Participants) | 15 | 8
  ISG15, Dose 4: Day 1 | 3.35 (5.212) | 1.24 (0.343)
  ISG15, Dose 4: Day 2: number analyzed (Participants) | 16 | 8
  ISG15, Dose 4: Day 2 | 19.09 (15.113) | 8.41 (20.782)
  ISG15, Dose 10: Day 1: number analyzed (Participants) | 15 | 8
  ISG15, Dose 10: Day 1 | 1.62 (0.742) | 1.02 (0.223)
  ISG15, Dose 10: Day 2: number analyzed (Participants) | 15 | 8
  ISG15, Dose 10: Day 2 | 19.71 (20.209) | 1.02 (0.366)
  ISG15, Early Study Drug Discontinuation: number analyzed (Participants) | 1 | 0
  ISG15, Early Study Drug Discontinuation | 1.14 |
  OAS-1, Dose 1: Day 2 | 6.83 (4.225) | 1.07 (0.285)
  OAS-1, Dose 4: Day 1: number analyzed (Participants) | 15 | 8
  OAS-1, Dose 4: Day 1 | 2.21 (2.087) | 1.13 (0.395)
  OAS-1, Dose 4: Day 2: number analyzed (Participants) | 16 | 8
  OAS-1, Dose 4: Day 2 | 7.44 (4.650) | 2.62 (4.676)
  OAS-1, Dose 10: Day 1: number analyzed (Participants) | 15 | 8
  OAS-1, Dose 10: Day 1 | 1.47 (0.665) | 1.03 (0.218)
  OAS-1, Dose 10: Day 2: number analyzed (Participants) | 15 | 8
  OAS-1, Dose 10: Day 2 | 6.83 (5.189) | 1.04 (0.162)
  OAS-1, Early Study Drug Discontinuation: number analyzed (Participants) | 1 | 0
  OAS-1, Early Study Drug Discontinuation | 1.08 |
  MX1, Dose 1: Day 2 | 9.36 (6.873) | 1.06 (0.249)
  MX1, Dose 4: Day 1: number analyzed (Participants) | 15 | 8
  MX1, Dose 4: Day 1 | 2.98 (4.650) | 1.17 (0.312)
  MX1, Dose 4: Day 2: number analyzed (Participants) | 16 | 8
  MX1, Dose 4: Day 2 | 9.91 (8.061) | 3.49 (6.957)
  MX1, Dose 10: Day 1: number analyzed (Participants) | 15 | 8
  MX1, Dose 10: Day 1 | 1.59 (0.844) | 1.03 (0.226)
  MX1, Dose 10: Day 2: number analyzed (Participants) | 15 | 8
  MX1, Dose 10: Day 2 | 10.29 (8.862) | 0.98 (0.232)
  MX1, Early Study Drug Discontinuation: number analyzed (Participants) | 1 | 0
  MX1, Early Study Drug Discontinuation | 1.06 |
Statistical Analysis 1: Comparison: Vesatolimod vs Placebo; ISG15, Dose 1: Day 2; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 2: Comparison: Vesatolimod vs Placebo; ISG15, Dose 4: Day 1; Test type: Superiority; p = 0.58, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 3: Comparison: Vesatolimod vs Placebo; ISG15, Dose 4: Day 2; Test type: Superiority; p = 0.009, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 4: Comparison: Vesatolimod vs Placebo; Test type: Superiority — ISG15, Dose 10: Day 1; p = 0.031, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 5: Comparison: Vesatolimod vs Placebo; ISG15, Dose 10: Day 2; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 6: Comparison: Vesatolimod vs Placebo; OAS-1, Dose 1: Day 2; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 7: Comparison: Vesatolimod vs Placebo; OAS-1, Dose 4: Day 1; Test type: Superiority; p = 0.057, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 8: Comparison: Vesatolimod vs Placebo; OAS-1, Dose 4: Day 2; Test type: Superiority; p = 0.009, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 9: Comparison: Vesatolimod vs Placebo; OAS-1, Dose 10: Day 1; Test type: Superiority; p = 0.057, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 10: Comparison: Vesatolimod vs Placebo; OAS-1, Dose 10: Day 2; Test type: Superiority; p = 0.005, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 11: Comparison: Vesatolimod vs Placebo; MX1, Dose 1: Day 2; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 12: Comparison: Vesatolimod vs Placebo; MX1, Dose 4: Day 1; Test type: Superiority; p = 0.17, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 13: Comparison: Vesatolimod vs Placebo; MX1, Dose 4: Day 2; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 14: Comparison: Vesatolimod vs Placebo; Test type: Superiority — MX1, Dose 10: Day 1; p = 0.100, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 15: Comparison: Vesatolimod vs Placebo; MX1, Dose 10: Day 2; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests

8. Secondary Outcome: Change From Baseline in Immune Cell Activation
Description: Activation of Immune cells (T cells: CD4/CD38/HLADR, CD8/CD38/HLADR and NK cells: CD69+CD56+CD16+, CD69+CD56dimCD16neg, CD69+CD56brCD16dim) was measured by cytometry.
Time Frame: Baseline and Dose 4: Days 1,2,4; Dose 6: Days 1,4; Dose 10: Days 1,2,4,14; ATI Remission Visit (12 weeks post ATI Visit: evaluated at maximum of 24 weeks)
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of cell activation
Arm/Group | Vesatolimod | Placebo
Number analyzed (Participants) | 9 | 6
percentage of cell activation
  CD4/CD38/HLADR, Baseline: number analyzed (Participants) | 8 | 6
  CD4/CD38/HLADR, Baseline | 2.7 (0.94) | 2.3 (1.04)
  CD4/CD38/HLADR,Change at Dose 4: Day 1: number analyzed (Participants) | 5 | 6
  CD4/CD38/HLADR,Change at Dose 4: Day 1 | 0.4 (0.58) | -0.3 (0.38)
  CD4/CD38/HLADR,Change at Dose 4: Day 2: number analyzed (Participants) | 5 | 6
  CD4/CD38/HLADR,Change at Dose 4: Day 2 | 0.9 (0.88) | 0.4 (1.02)
  CD4/CD38/HLADR,Change at Dose 4: Day 4: number analyzed (Participants) | 4 | 5
  CD4/CD38/HLADR,Change at Dose 4: Day 4 | 0.7 (0.53) | -0.3 (0.74)
  CD4/CD38/HLADR,Change at Dose 6: Day 1: number analyzed (Participants) | 4 | 6
  CD4/CD38/HLADR,Change at Dose 6: Day 1 | 0.5 (0.41) | -0.2 (0.90)
  CD4/CD38/HLADR,Change at Dose 6: Day 4: number analyzed (Participants) | 4 | 6
  CD4/CD38/HLADR,Change at Dose 6: Day 4 | 0.9 (0.41) | -0.1 (1.20)
  CD4/CD38/HLADR,Change at Dose 10: Day 1: number analyzed (Participants) | 3 | 5
  CD4/CD38/HLADR,Change at Dose 10: Day 1 | 1.0 (0.56) | -0.4 (0.45)
  CD4/CD38/HLADR,Change at Dose 10: Day 2: number analyzed (Participants) | 2 | 5
  CD4/CD38/HLADR,Change at Dose 10: Day 2 | 2.6 (0.11) | -0.3 (0.75)
  CD4/CD38/HLADR,Change at Dose 10: Day 4: number analyzed (Participants) | 4 | 6
  CD4/CD38/HLADR,Change at Dose 10: Day 4 | 1.0 (1.60) | -0.2 (1.45)
  CD4/CD38/HLADR,Change at Dose 10: Day 14: number analyzed (Participants) | 7 | 6
  CD4/CD38/HLADR,Change at Dose 10: Day 14 | 0.5 (0.36) | 0.1 (1.16)
  CD4/CD38/HLADR,Change at ATI Remission: number analyzed (Participants) | 0 | 2
  CD4/CD38/HLADR,Change at ATI Remission |  | 1.3 (1.63)
  CD8/CD38/HLADR, Baseline: number analyzed (Participants) | 8 | 6
  CD8/CD38/HLADR, Baseline | 5.4 (2.43) | 5.2 (2.86)
  CD8/CD38/HLADR,Change at Dose 4: Day 1: number analyzed (Participants) | 5 | 6
  CD8/CD38/HLADR,Change at Dose 4: Day 1 | 0.6 (1.41) | -0.8 (1.23)
  CD8/CD38/HLADR,Change at Dose 4: Day 2: number analyzed (Participants) | 5 | 6
  CD8/CD38/HLADR,Change at Dose 4: Day 2 | 1.6 (1.19) | 0.2 (2.06)
  CD8/CD38/HLADR,Change at Dose 4: Day 4: number analyzed (Participants) | 4 | 5
  CD8/CD38/HLADR,Change at Dose 4: Day 4 | 0.8 (0.56) | -0.9 (1.83)
  CD8/CD38/HLADR,Change at Dose 6: Day 1: number analyzed (Participants) | 4 | 6
  CD8/CD38/HLADR,Change at Dose 6: Day 1 | -0.6 (0.70) | -1.1 (1.56)
  CD8/CD38/HLADR,Change at Dose 6: Day 4: number analyzed (Participants) | 4 | 6
  CD8/CD38/HLADR,Change at Dose 6: Day 4 | 1.5 (1.53) | -0.7 (2.14)
  CD8/CD38/HLADR,Change at Dose 10: Day 1: number analyzed (Participants) | 3 | 5
  CD8/CD38/HLADR,Change at Dose 10: Day 1 | 1.5 (2.82) | -1.3 (1.77)
  CD8/CD38/HLADR,Change at Dose 10: Day 2: number analyzed (Participants) | 2 | 5
  CD8/CD38/HLADR,Change at Dose 10: Day 2 | 7.0 (4.83) | -1.2 (2.09)
  CD8/CD38/HLADR,Change at Dose 10: Day 4: number analyzed (Participants) | 4 | 6
  CD8/CD38/HLADR,Change at Dose 10: Day 4 | 3.0 (3.25) | -1.3 (2.31)
  CD8/CD38/HLADR,Change at Dose 10: Day 14: number analyzed (Participants) | 7 | 6
  CD8/CD38/HLADR,Change at Dose 10: Day 14 | 1.6 (3.03) | 0.0 (2.81)
  CD8/CD38/HLADR,Change at ATI Remission Visit: number analyzed (Participants) | 0 | 2
  CD8/CD38/HLADR,Change at ATI Remission Visit |  | 6.0 (6.41)
  CD69+CD56+CD16+, Baseline | 7.5 (7.04) | 6.7 (6.31)
  CD69+CD56+CD16+,Change at Dose 4: Day 1: number analyzed (Participants) | 6 | 6
  CD69+CD56+CD16+,Change at Dose 4: Day 1 | -2.2 (5.43) | -0.4 (3.24)
  CD69+CD56+CD16+,Change at Dose 4: Day 2: number analyzed (Participants) | 6 | 6
  CD69+CD56+CD16+,Change at Dose 4: Day 2 | 4.5 (7.45) | 0.5 (2.81)
  CD69+CD56+CD16+,Change at Dose 4: Day 4: number analyzed (Participants) | 5 | 5
  CD69+CD56+CD16+,Change at Dose 4: Day 4 | 1.0 (3.04) | 0.0 (5.12)
  CD69+CD56+CD16+,Change at Dose 6: Day 1: number analyzed (Participants) | 4 | 6
  CD69+CD56+CD16+,Change at Dose 6: Day 1 | 0.2 (2.36) | 0.4 (4.32)
  CD69+CD56+CD16+,Change at Dose 6: Day 4: number analyzed (Participants) | 4 | 6
  CD69+CD56+CD16+,Change at Dose 6: Day 4 | 0.9 (0.95) | -1.5 (4.78)
  CD69+CD56+CD16+,Change at Dose 10: Day 1: number analyzed (Participants) | 3 | 5
  CD69+CD56+CD16+,Change at Dose 10: Day 1 | 0.5 (0.61) | -1.2 (4.67)
  CD69+CD56+CD16+,Change at Dose 10: Day 2: number analyzed (Participants) | 2 | 5
  CD69+CD56+CD16+,Change at Dose 10: Day 2 | 11.1 (2.72) | -2.2 (5.81)
  CD69+CD56+CD16+,Change at Dose 10: Day 4: number analyzed (Participants) | 4 | 6
  CD69+CD56+CD16+,Change at Dose 10: Day 4 | 1.7 (1.99) | -1.4 (5.10)
  CD69+CD56+CD16+,Change at Dose 10: Day 14: number analyzed (Participants) | 7 | 6
  CD69+CD56+CD16+,Change at Dose 10: Day 14 | 0.8 (6.77) | -0.4 (3.92)
  CD69+CD56+CD16+,Change at ATI Remission Visit: number analyzed (Participants) | 0 | 2
  CD69+CD56+CD16+,Change at ATI Remission Visit |  | -1.7 (1.34)
  CD69+CD56dimCD16neg, Baseline | 12.2 (6.41) | 11.3 (10.37)
  CD69+CD56dimCD16neg,Change at Dose 4: Day 1: number analyzed (Participants) | 6 | 6
  CD69+CD56dimCD16neg,Change at Dose 4: Day 1 | -1.8 (5.13) | -0.7 (2.72)
  CD69+CD56dimCD16neg,Change at Dose 4: Day 2: number analyzed (Participants) | 6 | 6
  CD69+CD56dimCD16neg,Change at Dose 4: Day 2 | 6.7 (4.95) | -0.8 (4.10)
  CD69+CD56dimCD16neg,Change at Dose 4: Day 4: number analyzed (Participants) | 5 | 5
  CD69+CD56dimCD16neg,Change at Dose 4: Day 4 | 1.9 (6.02) | -1.1 (6.50)
  CD69+CD56dimCD16neg,Change at Dose 6: Day 1: number analyzed (Participants) | 4 | 6
  CD69+CD56dimCD16neg,Change at Dose 6: Day 1 | -0.7 (5.36) | -3.0 (7.89)
  CD69+CD56dimCD16neg,Change at Dose 6: Day 4: number analyzed (Participants) | 4 | 6
  CD69+CD56dimCD16neg,Change at Dose 6: Day 4 | 2.6 (3.81) | -3.0 (7.00)
  CD69+CD56dimCD16neg,Change at Dose 10: Day 1: number analyzed (Participants) | 3 | 5
  CD69+CD56dimCD16neg,Change at Dose 10: Day 1 | -0.7 (5.15) | -3.7 (7.02)
  CD69+CD56dimCD16neg,Change at Dose 10: Day 2: number analyzed (Participants) | 2 | 5
  CD69+CD56dimCD16neg,Change at Dose 10: Day 2 | 23.9 (8.15) | -4.2 (7.94)
  CD69+CD56dimCD16neg,Change at Dose 10: Day 4: number analyzed (Participants) | 4 | 6
  CD69+CD56dimCD16neg,Change at Dose 10: Day 4 | 2.0 (2.55) | -2.0 (6.70)
  CD69+CD56dimCD16neg,Change at Dose 10: Day 14: number analyzed (Participants) | 7 | 6
  CD69+CD56dimCD16neg,Change at Dose 10: Day 14 | 1.6 (4.89) | -2.5 (8.49)
  CD69+CD56dimCD16neg,Change at Dose 10: ATI Remission: number analyzed (Participants) | 0 | 2
  CD69+CD56dimCD16neg,Change at Dose 10: ATI Remission |  | -7.3 (13.15)
  CD69+CD56brCD16dim, Baseline | 5.0 (2.68) | 2.6 (1.02)
  CD69+CD56brCD16dim,Change at Dose 4: Day 1: number analyzed (Participants) | 6 | 6
  CD69+CD56brCD16dim,Change at Dose 4: Day 1 | -1.5 (1.46) | -0.3 (1.89)
  CD69+CD56brCD16dim,Change at Dose 4: Day 2: number analyzed (Participants) | 6 | 6
  CD69+CD56brCD16dim,Change at Dose 4: Day 2 | 1.0 (2.98) | 0.6 (2.49)
  CD69+CD56brCD16dim,Change at Dose 4: Day 4: number analyzed (Participants) | 5 | 5
  CD69+CD56brCD16dim,Change at Dose 4: Day 4 | 0.9 (1.63) | 2.9 (2.13)
  CD69+CD56brCD16dim,Change at Dose 6: Day 1: number analyzed (Participants) | 4 | 6
  CD69+CD56brCD16dim,Change at Dose 6: Day 1 | 1.9 (2.09) | 1.5 (2.90)
  CD69+CD56brCD16dim,Change at Dose 6: Day 4: number analyzed (Participants) | 4 | 6
  CD69+CD56brCD16dim,Change at Dose 6: Day 4 | 6.2 (6.68) | 0.2 (1.72)
  CD69+CD56brCD16dim,Change at Dose 10: Day 1: number analyzed (Participants) | 3 | 5
  CD69+CD56brCD16dim,Change at Dose 10: Day 1 | 5.0 (7.00) | 1.3 (1.72)
  CD69+CD56brCD16dim,Change at Dose 10: Day 2: number analyzed (Participants) | 2 | 5
  CD69+CD56brCD16dim,Change at Dose 10: Day 2 | 17.2 (16.49) | 2.2 (5.08)
  CD69+CD56brCD16dim,Change at Dose 10: Day 4: number analyzed (Participants) | 4 | 6
  CD69+CD56brCD16dim,Change at Dose 10: Day 4 | 0.0 (1.46) | 3.3 (3.70)
  CD69+CD56brCD16dim,Change at Dose 10: Day 14: number analyzed (Participants) | 7 | 6
  CD69+CD56brCD16dim,Change at Dose 10: Day 14 | 2.7 (3.14) | 0.9 (2.93)
  CD69+CD56brCD16dim,Change at ATI Remission: number analyzed (Participants) | 0 | 2
  CD69+CD56brCD16dim,Change at ATI Remission |  | 0.2 (0.91)
Statistical Analysis 1: Comparison: Vesatolimod vs Placebo; CD4/CD38/HLADR, Baseline; Test type: Superiority; p = 0.7469, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 2: Comparison: Vesatolimod vs Placebo; CD4/CD38/HLADR, Dose 4: Day 1; Test type: Superiority; p = 0.1207, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 3: Comparison: Vesatolimod vs Placebo; CD4/CD38/HLADR, Dose 4: Day 2; Test type: Superiority; p = 0.4113, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 4: Comparison: Vesatolimod vs Placebo; CD4/CD38/HLADR, Dose 4: Day 4; Test type: Superiority; p = 0.1113, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 5: Comparison: Vesatolimod vs Placebo; CD4/CD38/HLADR, Dose 6: Day 1; Test type: Superiority; p = 0.2410, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 6: Comparison: Vesatolimod vs Placebo; CD4/CD38/HLADR, Dose 6: Day 4; Test type: Superiority; p = 0.1098, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 7: Comparison: Vesatolimod vs Placebo; CD4/CD38/HLADR, Dose 10: Day 1; Test type: Superiority; p = 0.0369, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 8: Comparison: Vesatolimod vs Placebo; CD4/CD38/HLADR, Dose 10: Day 2; Test type: Superiority; p = 0.0814, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 9: Comparison: Vesatolimod vs Placebo; CD4/CD38/HLADR, Dose 10: Day 4; Test type: Superiority; p = 0.1658, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 10: Comparison: Vesatolimod vs Placebo; CD4/CD38/HLADR, Dose 10: Day 14; Test type: Superiority; p = 0.9431, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 11: Comparison: Vesatolimod vs Placebo; CD8/CD38/HLADR, Baseline; Test type: Superiority; p = 0.6514, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 12: Comparison: Vesatolimod vs Placebo; CD8/CD38/HLADR, Dose 4: Day 1; Test type: Superiority; p = 0.0821, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 13: Comparison: Vesatolimod vs Placebo; CD8/CD38/HLADR, Dose 4: Day 2; Test type: Superiority; p = 0.2353, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 14: Comparison: Vesatolimod vs Placebo; CD8/CD38/HLADR, Dose 4: Day 4; Test type: Superiority; p = 0.1779, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 15: Comparison: Vesatolimod vs Placebo; CD8/CD38/HLADR, Dose 6: Day 1; Test type: Superiority; p = 0.7491, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 16: Comparison: Vesatolimod vs Placebo; CD8/CD38/HLADR, Dose 6: Day 4; Test type: Superiority; p = 0.0700, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 17: Comparison: Vesatolimod vs Placebo; CD8/CD38/HLADR, Dose 10: Day 1; Test type: Superiority; p = 0.3711, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 18: Comparison: Vesatolimod vs Placebo; CD8/CD38/HLADR, Dose 10: Day 2; Test type: Superiority; p = 0.0814, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 19: Comparison: Vesatolimod vs Placebo; CD8/CD38/HLADR, Dose 10: Day 4; Test type: Superiority; p = 0.0700, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 20: Comparison: Vesatolimod vs Placebo; CD8/CD38/HLADR, Dose 10: Day 14; Test type: Superiority; p = 0.8303, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 21: Comparison: Vesatolimod vs Placebo; CD69+CD56+CD16+, Baseline; Test type: Superiority; p = 0.9530, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 22: Comparison: Vesatolimod vs Placebo; CD69+CD56+CD16+, Dose 4: Day 1; Test type: Superiority; p = 0.1735, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 23: Comparison: Vesatolimod vs Placebo; CD69+CD56+CD16+, Dose 4: Day 2; Test type: Superiority; p = 0.2971, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 24: Comparison: Vesatolimod vs Placebo; CD69+CD56+CD16+, Dose 4: Day 4; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 25: Comparison: Vesatolimod vs Placebo; CD69+CD56+CD16+, Dose 6: Day 1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 26: Comparison: Vesatolimod vs Placebo; CD69+CD56+CD16+, Dose 6: Day 4; Test type: Superiority; p = 0.3374, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 27: Comparison: Vesatolimod vs Placebo; CD69+CD56+CD16+, Dose 10: Day 1; Test type: Superiority; p = 0.7656, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 28: Comparison: Vesatolimod vs Placebo; CD69+CD56+CD16+, Dose 10: Day 2; Test type: Superiority; p = 0.0814, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 29: Comparison: Vesatolimod vs Placebo; CD69+CD56+CD16+, Dose 10: Day 4; Test type: Superiority; p = 0.3374, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 30: Comparison: Vesatolimod vs Placebo; CD69+CD56+CD16+, Dose 10: Day 14; Test type: Superiority; p = 0.4320, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 31: Comparison: Vesatolimod vs Placebo; CD69+CD56dimCD16neg, Baseline; Test type: Superiority; p = 0.8597, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 32: Comparison: Vesatolimod vs Placebo; CD69+CD56dimCD16neg, Dose 4: Day 1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 33: Comparison: Vesatolimod vs Placebo; CD69+CD56dimCD16neg, Dose 4: Day 2; Test type: Superiority; p = 0.0306, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 34: Comparison: Vesatolimod vs Placebo; CD69+CD56dimCD16neg, Dose 4: Day 4; Test type: Superiority; p = 0.8345, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 35: Comparison: Vesatolimod vs Placebo; CD69+CD56dimCD16neg, Dose 6: Day 1; Test type: Superiority; p = 0.9151, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 36: Comparison: Vesatolimod vs Placebo; CD69+CD56dimCD16neg, Dose 6: Day 4; Test type: Superiority; p = 0.1098, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 37: Comparison: Vesatolimod vs Placebo; CD69+CD56dimCD16neg, Dose 10: Day 1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 38: Comparison: Vesatolimod vs Placebo; CD69+CD56dimCD16neg, Dose 10: Day 2; Test type: Superiority; p = 0.0814, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 39: Comparison: Vesatolimod vs Placebo; CD69+CD56dimCD16neg, Dose 10: Day 4; Test type: Superiority; p = 0.4555, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 40: Comparison: Vesatolimod vs Placebo; CD69+CD56dimCD16neg, Dose 10: Day 14; Test type: Superiority; p = 0.6171, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 41: Comparison: Vesatolimod vs Placebo; CD69+CD56brCD16dim, Baseline; Test type: Superiority; p = 0.0677, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 42: Comparison: Vesatolimod vs Placebo; CD69+CD56brCD16dim, Dose 4: Day 1; Test type: Superiority; p = 0.4712, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 43: Comparison: Vesatolimod vs Placebo; CD69+CD56brCD16dim, Dose 4: Day 2; Test type: Superiority; p = 0.6889, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 44: Comparison: Vesatolimod vs Placebo; CD69+CD56brCD16dim, Dose 4: Day 4; Test type: Superiority; p = 0.1437, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 45: Comparison: Vesatolimod vs Placebo; CD69+CD56brCD16dim, Dose 6: Day 1; Test type: Superiority; p = 0.7491, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 46: Comparison: Vesatolimod vs Placebo; CD69+CD56brCD16dim, Dose 6: Day 4; Test type: Superiority; p = 0.0700, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 47: Comparison: Vesatolimod vs Placebo; CD69+CD56brCD16dim, Dose 10: Day 1; Test type: Superiority; p = 0.7656, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 48: Comparison: Vesatolimod vs Placebo; CD69+CD56brCD16dim, Dose 10: Day 2; Test type: Superiority; p = 0.1752, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 49: Comparison: Vesatolimod vs Placebo; CD69+CD56brCD16dim, Dose 10: Day 4; Test type: Superiority; p = 0.0700, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests
Statistical Analysis 50: Comparison: Vesatolimod vs Placebo; Test type: Superiority — CD69+CD56brCD16dim, Dose 10: Day 14; p = 0.2246, Wilcoxon (Mann-Whitney); P-values are based on two-sided Wilcoxon rank sum tests

9. Secondary Outcome: Pharmacokinetic (PK) Parameter: Cmax of Vesatolimod
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: Pre-dose (≤ 5 minutes prior to dosing), 0.5, 1, 2, 4, 6, 8, 10, and 24 hours post dose at Dose 1-Day 1 visit.
Population: The vesatolimod PK Analysis Set included all participants who were randomized into the study, received at least 1 dose of active vesatolimod, and had at least 1 non-missing post baseline concentration value for vesatolimod. Per planned analysis this outcome measure was analyzed by actual treatment received (i.e. 'Vesatolimod').
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Vesatolimod
Number analyzed (Participants) | 17
pg/mL | 7149.6 (7662.17)

10. Secondary Outcome: PK Parameter: AUClast of Vesatolimod
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Time Frame: Pre-dose (≤ 5 minutes prior to dosing), 0.5, 1, 2, 4, 6, 8, 10, and 24 hours post dose at Dose 1-Day 1 visit.
Population: Participants in the vesatolimod PK Analysis Set were analyzed. Per planned analysis this outcome measure was analyzed by actual treatment received (i.e. 'Vesatolimod').
Measure: Mean (Standard Deviation); unit: hour*pg/ml
Arm/Group | Vesatolimod
Number analyzed (Participants) | 17
hour*pg/ml | 49323.5 (48542.34)

11. Secondary Outcome: PK Parameter: AUCinf of Vesatolimod
Description: AUCinf was defined as the concentration of drug extrapolated to infinite time.
Time Frame: Pre-dose (≤ 5 minutes prior to dosing), 0.5, 1, 2, 4, 6, 8, 10, and 24 hours post dose at Dose 1-Day 1 visit.
Population: Participants in the vesatolimod PK Analysis Set with available data were analyzed. Per planned analysis this outcome measure was analyzed by actual treatment received (i.e. 'Vesatolimod').
Measure: Mean (Standard Deviation); unit: hour*pg/mL
Arm/Group | Vesatolimod
Number analyzed (Participants) | 16
hour*pg/mL | 60040.3 (59280.72)

12. Secondary Outcome: PK Parameter: %AUCexp of Vesatolimod
Description: %AUCexp is defined as the percentage of AUC extrapolated between AUClast and AUCinf.
Time Frame: Pre-dose (≤ 5 minutes prior to dosing), 0.5, 1, 2, 4, 6, 8, 10, and 24 hours post dose at Dose 1-Day 1 visit.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percentage of AUC
Arm/Group | Vesatolimod
Number analyzed (Participants) | 16
Percentage of AUC | 22.4 (7.90)

13. Secondary Outcome: PK Parameter: Tmax of Vesatolimod
Description: Tmax is defined as the time (observed time point) of Cmax.
Time Frame: Pre-dose (≤ 5 minutes prior to dosing), 0.5, 1, 2, 4, 6, 8, 10, and 24 hours post dose at Dose 1-Day 1 visit.
Population: as for outcome 11
Measure: Median (Full Range); unit: hour
Arm/Group | Vesatolimod
Number analyzed (Participants) | 16
hour | 2.00 [0.50 to 6.00]

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days after permanent discontinuation of study drug (assessed maximum up to 33 months and 5 days)
Description: The Safety Analysis Set included all participants who were randomized and received at least 1 dose of study drug.
Arm/Group | Vesatolimod | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/8
Other Adverse Events (participants affected / at risk) | 16/17 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vesatolimod (N=17) | Placebo (N=8)
Chronic gastritis (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vesatolimod (N=17) | Placebo (N=8)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Blepharospasm (Eye disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Angular cheilitis (Gastrointestinal disorders) | 1 | 0
Chapped lips (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Faeces soft (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 1
Swollen tongue (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 4 | 0
Fatigue (General disorders) | 3 | 0
Malaise (General disorders) | 2 | 0
Pyrexia (General disorders) | 3 | 0
Vessel puncture site bruise (General disorders) | 2 | 0
Acute sinusitis (Infections and infestations) | 2 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1
Laryngitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 3 | 2
Tinea cruris (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 5 | 3
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Morning sickness (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Haematospermia (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT03060447/SAP_000.pdf
  • Study Protocol (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT03060447/Prot_001.pdf